CLINICAL TRIAL: NCT06923670
Title: Prevalence Of Germline Gene Mutations In Patients With Myeloproliferative Neoplasms With Family History
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, CHIUSOLO PATRIZIA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 7221
Record Dates: First submitted 2025-03-26; First posted 2025-04-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Polycythemia Vera; Essential Thrombocythaemia; Myelofibrosis
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis | interventions — Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with familial history of hematological malignancies (Experimental): The investigators will evaluate the presence of mutations in the following genes: ABRAXAS1, ACD, ANKRD26, APC, ATG2B, ATM, BARD1, BMPR1A, BRCA1/2, BRIP1, CDH1, CDKN2A, CEBPA, CHECK2, CSF3R, DDX41, EPCAM, ERCC6L2, ETV6, FANCA, FANCB, FANCC, FANCD1, FANCD2, FANCE, FANCF, FANCG, FANCL, GATA2, GSKIP, MBD4, MECOM, MEN1, MLH1, MLH3, MRE11, MSH2, MSH6, MUTYH, NBN, NF1, NF2, PALB2, PIK3CA, POLD1, POLE, PMS2, PMS2CL, PTEN, PTPN11, RAD50, RAD51C, RAD51D, RET, RTEL1, RUNX1, SAMD9, SAMD9L, SBDS, SRP72, STK11, TERC, TERT, TP53, TSC1, TSC2, VHL, WAS, XRCC2
  Interventions: Diagnostic Test: NGS testing; Diagnostic Test: NGS analysis for mutations in genes involved in familial predisposition to hematological malignancies
- Patients without familial history of hematological malignancies (Active Comparator): The investigators will evaluate the presence of mutations in the following genes: ABRAXAS1, ACD, ANKRD26, APC, ATG2B, ATM, BARD1, BMPR1A, BRCA1/2, BRIP1, CDH1, CDKN2A, CEBPA, CHECK2, CSF3R, DDX41, EPCAM, ERCC6L2, ETV6, FANCA, FANCB, FANCC, FANCD1, FANCD2, FANCE, FANCF, FANCG, FANCL, GATA2, GSKIP, MBD4, MECOM, MEN1, MLH1, MLH3, MRE11, MSH2, MSH6, MUTYH, NBN, NF1, NF2, PALB2, PIK3CA, POLD1, POLE, PMS2, PMS2CL, PTEN, PTPN11, RAD50, RAD51C, RAD51D, RET, RTEL1, RUNX1, SAMD9, SAMD9L, SBDS, SRP72, STK11, TERC, TERT, TP53, TSC1, TSC2, VHL, WAS, XRCC2
  Interventions: Diagnostic Test: NGS testing; Diagnostic Test: NGS analysis for mutations in genes involved in familial predisposition to hematological malignancies

INTERVENTIONS:
Diagnostic Test: NGS testing — The investigators will test in NGS the presence of mutations in the following genes: ABRAXAS1, ACD, ANKRD26, APC, ATG2B, ATM, BARD1, BMPR1A, BRCA1/2, BRIP1, CDH1, CDKN2A, CEBPA, CHECK2, CSF3R, DDX41, EPCAM, ERCC6L2, ETV6, FANCA, FANCB, FANCC, FANCD1, FANCD2, FANCE, FANCF, FANCG, FANCL, GATA2, GSKIP, MBD4, MECOM, MEN1, MLH1, MLH3, MRE11, MSH2, MSH6, MUTYH, NBN, NF1, NF2, PALB2, PIK3CA, POLD1, POLE, PMS2, PMS2CL, PTEN, PTPN11, RAD50, RAD51C, RAD51D, RET, RTEL1, RUNX1, SAMD9, SAMD9L, SBDS, SRP72, STK11, TERC, TERT, TP53, TSC1, TSC2, VHL, WAS, XRCC2
Diagnostic Test: NGS analysis for mutations in genes involved in familial predisposition to hematological malignancies — The investigators will evaluate the presence of mutations in the following genes: ABRAXAS1, ACD, ANKRD26, APC, ATG2B, ATM, BARD1, BMPR1A, BRCA1/2, BRIP1, CDH1, CDKN2A, CEBPA, CHECK2, CSF3R, DDX41, EPCAM, ERCC6L2, ETV6, FANCA, FANCB, FANCC, FANCD1, FANCD2, FANCE, FANCF, FANCG, FANCL, GATA2, GSKIP, MBD4, MECOM, MEN1, MLH1, MLH3, MRE11, MSH2, MSH6, MUTYH, NBN, NF1, NF2, PALB2, PIK3CA, POLD1, POLE, PMS2, PMS2CL, PTEN, PTPN11, RAD50, RAD51C, RAD51D, RET, RTEL1, RUNX1, SAMD9, SAMD9L, SBDS, SRP72, STK11, TERC, TERT, TP53, TSC1, TSC2, VHL, WAS, XRCC2

SUMMARY:
Philadelphia-negative myeloproliferative neoplasms (MPNs) occur sporadically and are due to somatic mutations in the JAK2 (Janus kinase 2), CALR (calreticulin) and MPL (thrombopoietin receptor) genes. However, data from epidemiological and family studies clearly highlight a heritable component that influences the risk of developing MPN and potentially contributes to the observed phenotypic pleiotropy. Genome-wide association studies in MPN familial clusters have identified a number of germline genetic variants associated with an increased risk of developing MPN. The strongest association discovered so far is the presence of the JAK2 46/1 haplotype and, subsequently, several studies have found additional variants in other genes, particularly in the TERT gene.

The aim of the study would be to investigate the presence of germline mutations in MPN patients selected on the basis of a family history of myeloid neoplasms through the analysis of both already recognized genes and other potentially implicated ones.

ELIGIBILITY:
Inclusion Criteria:

*Patients >18 years

* Diagnosis of MPN (Essential Thrombocythemia, Polycythemia Vera, Myelofibrosis) confirmed according to ICC 2022 criteria
* Familiarity for myeloid neoplasia: at least one first or second degree relative affected by myeloid neoplasia (probands) OR presence of matching criteria with a proband (controls). Each center will be able to contribute with its own available patients/relatives, providing the clinical-laboratory data required by the study.

  * Signing of informed consent according to ICH/EU/GCP and local national laws (if applicable)

Exclusion Criteria:

* Patients <18 years Patients with other hematological diagnoses; • Lack of informed consen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2025-05-21 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between clinical characteristis in patients with and without family history: | 30 months
  Complete blood count test Presence of splenomegaly Presence of Fibrosis at bone marrow biopsy
Comparison between biological characteristis in patients with and without family history: | 30 months
  Presence of driver mutations:
  JAK2 V617F Calreticulin mutations MPL mutations
  Presence of detrimental mutations in the following genes: ASXL1, ZSFR2, IDH1, IDH2, EZH2, TP53

SECONDARY OUTCOMES:
Prevalence of germline mutations in MPN patients | 36 months
  Prevalence of germline mutations in MPN patients with familial hystory in the following genes:
  ABRAXAS1, ACD, ANKRD26, APC, ATG2B, ATM, BARD1, BMPR1A, BRCA1/2, BRIP1, CDH1, CDKN2A, CEBPA, CHECK2, CSF3R, DDX41, EPCAM, ERCC6L2, ETV6, FANCA, FANCB, FANCC, FANCD1, FANCD2, FANCE, FANCF, FANCG, FANCL, GATA2, GSKIP, MBD4, MECOM, MEN1, MLH1, MLH3, MRE11, MSH2, MSH6, MUTYH, NBN, NF1, NF2, PALB2, PIK3CA, POLD1, POLE, PMS2, PMS2CL, PTEN, PTPN11, RAD50, RAD51C, RAD51D, RET, RTEL1, RUNX1, SAMD9, SAMD9L, SBDS, SRP72, STK11, TERC, TERT, TP53, TSC1, TSC2, VHL, WAS, XRCC2
Distribution of hematologic malignancies in the group with familial hystory | 36
  Prevalence of hematological malignancies in the group with familial history

IPD SHARING:
Plan to Share IPD: Undecided